CLINICAL TRIAL: NCT00172588
Title: Evaluation of Endometrial Stromal Cell Apoptosis in Adenomyosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361701197
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-11-28 (Estimated); Status verified 2004-12

CONDITIONS: Endometriosis
Keywords: adenomyosis; apoptosis; flowcytometry
MeSH Terms: conditions — Endometriosis; Adenomyosis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Our previous results revealed that the expression of killer inhibitory receptors (KIRs) on NK cells was decreased in eutopic endometrium in women with adenomyosis. It implies that the formation of adenomyosis might be due to abnormal endometrial tissues, but not the aberrant local immunological dysfunction in myometrium. In addition, in vitro coculture of macrophages and endometrial stromal cells (ESC) increase the expression of IL-6 mRNA in ESC, which might further enhance the proliferation of ESC and subsequently result in the formation of ectopic endometrial implants in adenomyosis. Besides, another possible mechanism is the abnormal apoptosis of ESC in adenomyosis. In endometriosis, apoptotic endometrial cells were found to be decreased, which possibly accounts for the formation of endometriosis. However, there have not been reports investigating the apoptosis of ESC in adenomyosis.

In this study, we try to investigate apoptotic ESC with flow cytometry in women with and without adenomyosis. Annexin V, bcl-2, and caspase-3 were measured to represent the degree of apoptosis in ESC.

DETAILED DESCRIPTION:
Eutopic endometrium was obtained and separated into single endometrial stromal cell (ESC) in women with adenomyosis (study group) and without adenomyosis (control group).

Annexin V-PE, bcl-2-PE, and caspase-3-PE are stained, and flow cytometry is done to measure the degree of apoptosis in ESC. On the other hand, another half of ESC are cultured for 24h, and also Annexin V-PE, bcl-2-PE, and caspase-3-PE are stained, and flow cytometry is done.

ELIGIBILITY:
Inclusion Criteria:

* women with adenomyosis
* at early- to mid-secretory phases

Exclusion Criteria:

* postmenopausal
* malignancy

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40
Dates: Start 2005-01; Study Completion 2005-10

CONTACTS AND LOCATIONS:
Overall Officials: Jehn-Hsiahn Yang, M.D., Principal Investigator — Department of Obstetrics and Gynecology, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan